CLINICAL TRIAL: NCT03675178
Title: Anerning Particle for Reducing the Application of Antibiotics of Childhood Community-acquired Pneumonia: a Randomized, Double Blind, Control of Placebo, Multi-center Clinical Study
Brief Title: Clinical Study of Anerning Particle for the Treatment of Childhood Community-acquired Pneumonia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Collaborators: The First Affiliated Hospital of Tianjin University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Yanming Xie, Deputy director, China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Anerning particle
Record Dates: First submitted 2018-08-05; First posted 2018-09-18 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Community-acquired Pneumonia
Keywords: Anerning particle; Clinical endpoint antibiotic application frequency; efficacy and safety; randomized; double blind
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Ceftriaxone; Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): Anerning particle +ceftriaxone sodium
  Interventions: Drug: Anerning particle
- control group (Placebo Comparator): Anerning particle placebo+ceftriaxone sodium
  Interventions: Drug: control group

INTERVENTIONS:
Drug: Anerning particle — Anerning particle ,1 bag/time,3 times/ day, +ceftriaxone sodium,50mg/kg/time, 1 time/day, the total amount per day does not exceed 2g，for 10 days.When the condition is cured, stop the medicine at any time.
  Other Names: ceftriaxone sodium
  Arms: treatment group
Drug: control group — Anerning particle placebo ,1 bag/time,3 times/ day, +ceftriaxone sodium,50mg/kg/time, 1 time/day, the total amount per day does not exceed 2g，for 10 days.When the condition is cured, stop the medicine at any time.
  Other Names: Anerning particle placebo
  Arms: control group

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and whether it can reduction of antibiotic use in the treatment of community-acquired pneumonia in children with Anerning granules combined with ceftriaxone sodium.

DETAILED DESCRIPTION:
To evaluate the efficacy, safety and whether it can reduction of antibiotic use in the treatment of community-acquired pneumonia in children with Anerning granules combined with ceftriaxone sodium.In this study, a randomized, double blind, parallel control of placebo, multi-center clinical study will be established. According to the relevant regulations of the CFDA, 216 cases need to be registered at least.The aim population is children who suffering of community-acquired pneumonia from September 2018 to December 2019. These cases will be devided into treatment group（Anerning particle+ Intravenous ceftriaxone sodium）,control group（Anerning particle simulants+ Intravenous ceftriaxone sodium）. Each group will be treated for 10 days hospitalization and if there is adverse drug reaction during treatment, follow-up until the laboratory indicators are normal. The efficacy indicators of this study were mainly from three dimensions: Frequency of antibiotics at the clinical endpoint, Total disease efficiency, Clinical recovery time. The symptom scores changes of each group before and after treatment were observed.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for children's CAP Western medicine and consider bacterial infection;
2. Those who meet the diagnostic criteria of TCM syndrome differentiation of wind-heat and closed lung syndrome;
3. Children aged 1 to 5 years old;
4. Within 48 hours of onset of CAP;
5. The informed consent process is in compliance with the regulations, and the legal representative signs the informed consent form.

Exclusion Criteria:

1. Chest X-ray films showed obvious lung tumors and tuberculosis;
2. Those with acute infectious diseases such as measles, whooping cough, and influenza;
3. Other upper respiratory tract infections, wheezing-like bronchitis, bronchial asthma, bronchial foreign bodies and other respiratory diseases;
4. Children with severe malnutrition and immunodeficiency;
5. Combine severe primary diseases such as severe heart, liver, kidney, digestion and hematopoietic system;
6. Those who meet the CAP (severe) Western diagnostic criteria for children;
7. Clinically diagnosed or clinically considered viral pneumonia, Mycoplasma pneumoniae pneumonia;
8. allergic constitution (allergic to more than 2 types of substances), or allergic to penicillins, cephalosporin antibiotics and Anering granules and their components;
9. Researchers believe that it is not appropriate to join the group.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 216 (Estimated)
Dates: Start 2018-09-22 (Estimated); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Whether Anerning particle can reduce the use of antibiotics | After 10 days of medication.When the condition is cured, stop the medicine at any time.
  Frequency of antibiotics (DDDs) at clinical endpoints of the two groups

SECONDARY OUTCOMES:
The chest X-ray of 216 participants will be assessed. | The maximum time for administration according to the protocol is 10 days, and the drug can be stopped at any time during clinical cure. If it is not good to change on the 6th day of treatment, use other measures.
  If the chest radiograph returns to normal, it indicates that the patient has recovered.
The blood routine and c-reactive protein of 216 participants will be assessed. | The maximum time for administration according to the protocol is 10 days, and the drug can be stopped at any time during clinical cure. If it is not good to change on the 6th day of treatment, use other measures.
  Combined detection of c-reactive protein and white blood cell， if the two indicators return to normal after treatment, the child recovers.
Complete fever time | The maximum time for administration according to the protocol is 10 days, and the drug can be stopped at any time during clinical cure. If it is not good to change on the 6th day of treatment, use other measures.
  Judging criteria: body temperature (underarm temperature) <37.3 ° C, and maintained for 24h and above. Measurement method: measured every 8h.

CONTACTS AND LOCATIONS:
Overall Officials: Yanming Xie, BA, Principal Investigator — Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences

IPD SHARING:
Plan to Share IPD: No